CLINICAL TRIAL: NCT06104332
Title: Post-marketing Clinical Investigation to Assess Real-life Usage Effectiveness, Safety and Patient Satisfaction of a Range of Hypertonic Seawater-based Decongestant Nasal Sprays
Brief Title: PMCF to Assess Real-life Usage Effectiveness, Safety and Patient Satisfaction of a Range of Hypertonic Seawater-based Decongestant Nasal Sprays
Status: Completed | Type: Observational
Sponsor: Laboratoire de la Mer (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Other Study IDs: PMCF Hyper Mini
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Allergic Rhinitis; URTI
Keywords: Medical device; Hypertonic seawater-based nasal spray
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- ProRhinel Naturel spray nasal/ Allergic Rhinitis
  Interventions: Device: ProRhinel Naturel spray nasal/ Allergic rhinitis
- ProRhinel Naturel spray nasal/ URTI
  Interventions: Device: ProRhinel Naturel spray nasal/ URTI
- ProRhinel EXTRA Eucalyptus spray nasal/ URTI
  Interventions: Device: ProRhinel EXTRA Eucalyptus spray nasal
- RESPIMER Enfant/ URTI
  Interventions: Device: RESPIMER Enfant
- Phytosun Aroms spray nasal MAX/ URTI
  Interventions: Device: Phytosun Aroms spray nasal MAX
- PHYSIOMER RHUME TRIPLE ACTION/ URTI
  Interventions: Device: PHYSIOMER RHUME TRIPLE ACTION
- Phytosun Aroms spray nasal decongestionnant/ URTI
  Interventions: Device: Phytosun Aroms spray nasal decongestionnant

INTERVENTIONS:
Device: ProRhinel Naturel spray nasal/ Allergic rhinitis — ProRhinel Naturel spray nasal: 21 days; 1 spray per nostril; 3 to 6 times per day
  Groups: ProRhinel Naturel spray nasal/ Allergic Rhinitis
Device: ProRhinel EXTRA Eucalyptus spray nasal — ProRhinel EXTRA Eucalyptus spray nasal: until resolution of symptoms (period of 14 days maximum) ; 2 to 3 sprays per nostril; 6 times per day maximum
  Groups: ProRhinel EXTRA Eucalyptus spray nasal/ URTI
Device: RESPIMER Enfant — RESPIMER Enfant: until resolution of symptoms (period of 14 days maximum) ; 1 spray per nostril; 4 times per day maximum
  Groups: RESPIMER Enfant/ URTI
Device: Phytosun Aroms spray nasal MAX — Phytosun Aroms spray nasal MAX: until resolution of symptoms (period of 14 days maximum) ; 1 spray per nostril; up to 4-6 times per day
  Groups: Phytosun Aroms spray nasal MAX/ URTI
Device: PHYSIOMER RHUME TRIPLE ACTION — PHYSIOMER RHUME TRIPLE ACTION: until resolution of symptoms (period of 14 days maximum) ; 1 spray per nostril; up to 4-6 times per day
  Groups: PHYSIOMER RHUME TRIPLE ACTION/ URTI
Device: Phytosun Aroms spray nasal decongestionnant — Phytosun Aroms spray nasal decongestionnant : until resolution of symptoms (period of 14 days maximum) ; 1 spray per nostril; 6 times per day maximum
  Groups: Phytosun Aroms spray nasal decongestionnant/ URTI
Device: ProRhinel Naturel spray nasal/ URTI — ProRhinel Naturel spray nasal: until resolution of symptoms (period of 14 days maximum) ; 1 spray per nostril; 3 to 6 times per day
  Groups: ProRhinel Naturel spray nasal/ URTI

SUMMARY:
The brief of this observational study is to evaluate usage, efficacy, safety and patient satisfaction of a range of hypertonic seawater-based decongestant nasal sprays in general population.

The main questions it aims to answer are:

* Usage,
* Efficacy,
* Safety,
* Satisfaction, in real-life usage with children, adults and pregnant or breastfeeding women. Participants will use the nasal spray as usual habits and complete daily questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Subject coming to pharmacy for spontaneous purchase of one of the medical device under investigation.
* Subject willing to buy one of the medical device under investigation following advice from pharmacist, general practitioner or any other health care professionals.
* Adult and children from 3 years old in compliance with the information for use.
* Subject presenting moderate nasal congestion or more.
* Subject agreeing to follow the study requirements during the whole study period.
* Subject having daily access to internet in order to answer online questionnaire.
* Subject able to understand verbal and written local language and in capacity to fill-in questionnaire himself.
* Subject able to give inform consent.

Exclusion Criteria:

* Subject with contraindications according to the information for use.
* Hypersensitivity or know allergy to any component of the product.
* Subject taking part in another clinical study or being in the exclusion period of another clinical study.
* Subject already included once in this study or having a family member already included in this study for the same indication.
* Vulnerable subject (except children, pregnant and breastfeeding women).

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General population coming to pharmacy for spontaneous purchase of a hypertonic seawater-based decongestant nasal spray for URTI or allergic rhinitis.
Sampling Method: Non-Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2023-11-04 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
URTI population : Effectiveness to improve nasal congestion | URTI: 3 days
  URTI: Assess effectiveness to improve nasal congestion in real world usage (6-point Likert scale) 6-point-Likert scale: 0 (None) - 1 (Very mild) - 2 (Mild) - 3 (Moderate) - 4 (Strong) - 5 (Very strong). Higher score means a worse outcome
AR population: Effectiveness to improve nasal congestion | AR: 7 days
  Allergic Rhinitis (AR) : Assess effectiveness to improve nasal congestion in real world usage (6-point Likert scale) 6-point-Likert scale: 0 (None) - 1 (Very mild) - 2 (Mild) - 3 (Moderate) - 4 (Strong) - 5 (Very strong). Higher score means a worse outcome

SECONDARY OUTCOMES:
Effectiveness to improve overall nasal symptoms (daytime) | URTI: Day 0 - Day 14
  URTI: Assess effectiveness (daytime) to improve overall nasal symptoms in real world usage (6-point Likert scale)
Effectiveness to improve overall nasal symptoms (daytime) | AR: Day 0 - Day 21
  AR: Assess effectiveness (daytime) to improve overall nasal symptoms in real world usage (6-point Likert scale)
Effectiveness to improve overall nasal symptoms (night-time) | URTI: Day 0 - Day 14
  URTI: Assess effectiveness (night-time) to improve overall nasal symptoms in real world usage (6-point Likert scale)
Effectiveness to improve overall nasal symptoms (night-time) | AR: Day 0 - Day 21
  AR: Assess effectiveness (night-time) to improve overall nasal symptoms in real world usage
Effectiveness to improve quality of life | URTI: Day 0 - Day 14
  URTI: Assess effectiveness to improve quality of life in real world usage (RQLQ self-administered questionnaire)
Effectiveness to improve quality of life | AR: Day 0 - Day 21
  AR: Assess effectiveness to improve quality of life in real world usage (RQLQ self-administered questionnaire)
Relief of nasal symptoms | AR: Day 1 - Day 21
  AR : assessment of nasal symptoms relief (7-point Likert scale)
Relief of nasal symptoms | URTI: Day 1 - Day 14
  URTI: assessment of nasal symptoms relief (7-point Likert scale)
Onset of action & Duration | URTI: Day 0 - Day 14
  URTI: Assess Onset of action & Duration (2 closed questions)
Onset of action & Duration | AR: Day 0 - Day 21
  AR: Assess Onset of action & Duration (2 closed questions)
Safety of the medical device | URTI: Day 0 - Day 14
  URTI: occurence of incidents and deficiencies
Tolerance | URTI: Day 14
  URTI: 1 question (numeric scale : 0-10)
Safety of the medical device | AR: Day 0 - Day 21
  AR: occurence of incidents and deficiencies
Tolerance | AR: Day 10 + Day 21
  AR: 1 question (numeric scale: 0-10)
Usage | URTI: Day 0 - Day 14
  URTI: number of day of use, number of use/ day, number of puff/ nostril, moment of use
Usage | AR: Day 0 - Day 21
  AR: number of day of use, number of use/ day, number of puff/ nostril, moment of use
Patient satisfaction | URTI: Day 14
  URTI: 10 questions on Satisfaction (numeric scale: 0-10)
Patient satisfaction | AR: Day 10 + Day 21
  AR: 10 questions on Satisfaction (numeric scale: 0-10)
Sensory profile | URTI: Day 14
  URTI: 4 questions on sensory profile (numeric scale: 0-10)
Sensory profile | AR: Day 10 + Day 21
  AR: 4 questions on sensory profile (numeric scale: 0-10)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Alexandra Crevecoeur, Honfleur
  - Annie Le Gall, Vern-sur-Seiche

IPD SHARING:
Plan to Share IPD: No